CLINICAL TRIAL: NCT06429631
Title: The Effects of CIC Training With a Mobile Application on Quality of Life and Compliance in Spinal Cord Injury Patients: a Single Blind Randomized Controlled Study (CIC: Clean Intermittent Catheterization)
Brief Title: The Effects of CIC Training With a Mobile Application on Quality of Life and Compliance in Spinal Cord Injury Patients: a Single Blind Randomized Controlled Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziler Physical Medicine and Rehabilitation Education and Research Hospital (Other)
Collaborators: Gazi University (Other)
Responsible Party: Principal Investigator, Nilgün Aras, Nurse, RN, MSN, Phd, Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 77082166-302.08.01-424987
Record Dates: First submitted 2024-05-18; First posted 2024-05-28 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Neurogenic Bladder; Spinal Cord Injury; Intermittent Catheterization; Mobile Application
Keywords: neurogenic bladder; education; mobil application; compliance; quality of life
MeSH Terms: conditions — Urinary Bladder, Neurogenic; Spinal Cord Injuries; Patient Compliance

STUDY DESIGN:
Intervention Model Description: parallel group single-blind randomized control trial
Who Masked: Participant
Masking Description: The person doing the statistical analysis will not know which is the experiment and which is the control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group(routine CIC education) (No Intervention): This group has routine CIC education. They fill the scales before discharge and 12. week after discharge.
- experimental group(routine CIC education+mobile application on telephone) (Experimental): This group has routine CIC education. Also mobile application uploaded their telephone before discharge.
  They fill the scales before discharge and 12. week after discharge.
  Interventions: Device: mobile application on telephone

INTERVENTIONS:
Device: mobile application on telephone — when patient discharge from the hospital, mobile application downloaded their telephone. then researcher give feedback about patients CIC outputs.
  also mobile application include 2 animations, videos, "frequently asked questions" and "ask the expert" section.
  Arms: experimental group(routine CIC education+mobile application on telephone)

SUMMARY:
Neurogenic bladder is a condition that occurs due to nerve damage or congenital problems and causes urination disorders. Nowadays, in individuals diagnosed with neurogenic bladder, Clean Intermittent Catheterization is often used to evacuate the urine accumulated in the bladder. Clean Intermittent Catheterization(CIC) is a simple, safe and effective method in which the catheter is placed through the meatus. In this application, the catheter is removed without waiting after urine drainage is achieved. This process is usually performed on its own. Since IC(Intermittent Catheterization) is a procedure performed on the bladder, it may cause some complications. IC application must be performed successfully to prevent or reduce complications. The success of the technique largely depends on patient education and follow-up. Sometimes patients may not be able to come to the hospital for follow-up and feedback after IC training.

Innovations are needed to ensure the continuation of distance education so that the education of patients who cannot come to the hospital is not incomplete. The literature includes brochures, videos, websites and some mobile applications for IC training. However, no application has been found that monitors patients' urine amounts.

This research was planned to examine the effect of clean intermittent catheterization training given via mobile application to individuals with spinal cord injury on their quality of life and compliance.

DETAILED DESCRIPTION:
scales:

1. Information form: Authors will ask to patients age, weight, height, gender, marital status, education level, diagnosis, time of injury, cause of injury, independence level, working or not working, presence of spasticity
2. WHOQOL-BREF(World Health Organization Quality of Life Scale):The WHO Quality of Life Assessment (WHOQOL) is a generic quality of life instrument that was designed to be applicable to people living under different circumstances, conditions, and cultures. The short version known as WHOQOL-BREF with 27 itemsin Turkish version. It is based on a Likert-type scale and is scored from 1 to 5, with higher scores indicating a better quality of life.
3. Intermittent Self-Catheterization Questionnaire (ISC-Q): This is a 24-item self-administered questionnaire. Each item is scored on a 5-point Likert-type scale ranging from 0 (strongly disagree) to 4 (strongly agree), and after the conversion of the 14 reverse-coded items to give a common range of 0-100, the scores are calculated by multiplying the mean value of all items within each domain by 25. The total ISC-Q score is then calculated from the simple average from across the four domains (0-100), with higher scores indicating a higher quality of life.
4. Intermittent Catheterization Adherence Scale (ICAS): ICAS (IntermittentCatheterization Adherence Scale) is used to assess long-term patient adherence to prescribed ISC treatment. Binary answers were used for the first seven questions:yes = 1, no = 0, whereas the response options for the eighth question were graded on a 5-point Likert-type scale: 0 indicating "never," 0.25 "sometimes," 0.5 "often,"0.75 "regularly," and 1 "always," leading to a maximum possible score of 8. A patient's score is empirically classified into three intervals: strong adherence = 0; average adherence = 1-2; low adherence = 3-8.
5. Mobile Application Usability Scale (MAUS): The scale measures mobile application usability which is formed with 10 constructs/factors which includes four items each (40 items at total). The scale measures using a 7-point Likert-type scale (1=strongly disagree…7=strongly agree)

ELIGIBILITY:
The study inclusion criteria were (1) 18-65 years of age, (2) receiving CIC training for the first time, (3) having sufficient manual dexterity, (4) using a single-use hydrophilic catheter, (5) having an IOS/Android phone and internet access, (6) having no vision problems, (7) having a Body Mass Index (BMI) <30, (8) speaking Turkish.

Participants were excluded if (1) they wanted to withdraw from the study, (2) they did not complete the data collection forms, (3) the doctor decided they should stop CIC, (4) they did not use the mobile application in the intervention group, and (5) they had received CIC training more than one month ago.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
1. WHOQOL-BREF(World Health Organization Quality of Life questionnaire), | Patients fill the scale "before discharge" and 12 weeks after discharge.
  This study want to evaluate quality of life with 2 scales. WHOQOL-BREF(World Health Organization Quality of Life Scale):The WHO Quality of Life Assessment (WHOQOL) is a generic quality of life instrument that was designed to be applicable to people living under different circumstances, conditions, and cultures. The short version known as WHOQOL-BREF with 26 items. Turkish version is 27 items. It is based on a Likert-type scale and is scored from 1 to 5, with higher scores indicating a better quality of life.
2. Intermittent Self-Catheterization Questionnaire (ISC-Q) | Patients fill the scale "before discharge" and 12 weeks after discharge.
  This is a 24-item self-administered questionnaire. Each item is scored on a 5-point Likert-type scale ranging from 0 (strongly disagree) to 4 (strongly agree), and after the conversion of the 14 reverse-coded items to give a common range of 0-100, the scores are calculated by multiplying the mean value of all items within each domain by 25. The total ISC-Q score is then calculated from the simple average from across the four domains (0-100), with higher scores indicating a higher quality of life.

SECONDARY OUTCOMES:
Intermittent Catheterization Adherence Scale (ICAS) | Patients fill the scale "before discharge" and 12 weeks after discharge.
  This study want to evaluate compliance with one scale. ICAS (IntermittentCatheterization Adherence Scale) is used to assess long-term patient adherence to prescribed ISC treatment. Binary answers were used for the first seven questions:yes = 1, no = 0, whereas the response options for the eighth question were graded on a 5-point Likert-type scale: 0 indicating "never," 0.25 "sometimes," 0.5 "often,"0.75 "regularly," and 1 "always," leading to a maximum possible score of 8. A patient's score is empirically classified in to three intervals: strong adherence = 0; average adherence = 1-2; low adherence = 3-8.

OTHER OUTCOMES:
Mobile Application Usability Scale (MAUS) | Only the experimental group completes this scale 12 weeks after discharge.
  The scale measures mobile application usability which is formed with 10 constructs/factors which includes four items each (40 items at total). The scale measures using a 7-point Likert-type scale (1=strongly disagree…7=strongly agree)

CONTACTS AND LOCATIONS:
Overall Officials: NURCAN ÇALIŞKAN, Prof. Dr, Principal Investigator — Gazi University; BİLGE YILMAZ, Prof. Dr., Principal Investigator — SBÜ GAZİLER FİZİK TEDAVİ VE REHABİLİTASYON EĞİTİM VE ARAŞTIRMA HASTANESİ; Nilgün Aras, Phd student, Study Chair — SBÜ GAZİLER FİZİK TEDAVİ VE REHABİLİTASYON EĞİTİM VE ARAŞTIRMA HASTANESİ
Locations (1):
- Ankara Gaziler Physical Therapy and Rehabilitation Training and Research Hospital, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Since the study is still not finished, it was decided not to share it.